CLINICAL TRIAL: NCT06053632
Title: The Effect of Eccentric Exercises on Lower Limb Muscle Imbalances and Functional Status of Young Female Football Players
Brief Title: Young Age Soccer Player's Lower Limb Muscle Imbalance and Functional Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LithuananianSportsU-15
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Young age soccer player; Eccentric hamstring exercise; Dynamic balance; Contractile muscle properties

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group will be asked to maintain their usual lifestyle.
- Experimental group (Experimental): The research group performed additional low-load and high-velocity - lying prone - eccentric hamstring exercise 3 times per week for 4 weeks. 12 sessions in total.
  Interventions: Behavioral: Low-load and high-velocity - lying prone - eccentric hamstring exercise

INTERVENTIONS:
Behavioral: Low-load and high-velocity - lying prone - eccentric hamstring exercise — Low-load and high-velocity - lying prone - eccentric hamstring exercise 3 times per week for 4 weeks.
  Arms: Experimental group

SUMMARY:
A randomized controlled trial is designed to examine the effects of low-load and high-velocity eccentric exercises on lower limb muscular properties, imbalances and functional status of 13-15 years old female football players.

DETAILED DESCRIPTION:
Twenty participants were included in the study. All participants were divided in two groups - control and experimental. In the experimental group (n=10) participants after team soccer training additional received 4 weeks eccentric exercises, in the control group (n=10) - did not perform additional exercises. The research group performed additional low-load and high-velocity - lying prone - eccentric hamstring exercise 3 times per week for 4 weeks. Pre- and post- training assessment included concentric/eccentric knee extension and flexion at 60°/s and 120°/s, changes in muscle contractile characteristics and dynamic balance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy players able to participate in training and competitions.
* Playing football for at least 2 years.
* Regularly participating in team training, 2-3 times a week.

Exclusion Criteria:

* Female soccer players with a lower extremity injury (in a period of 6 months)
* Pain is less than 2 points on the Visual Analog Pain Scale.
* Irregular exercise
* The number of years of training attended is too low

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in isokinetic peak torque (with Biodex) | Baseline and after 4 weeks
  Knee extension/flexion isokinetic peak torque measurements will be done at 60°/s, 120°/s
Dynamic balance | Baseline and after 4 weeks
  Y-balance Test evaluates lower extremity strength, knee stability and dynamic balance in anterior, posteromedial and posterolateral direction. For each direction, three practice trials were allowed before three test trials were recorded. Mean reach distances (cm) was normalized to leg length, which was measured from the anterior superior iliac spine to the most distal portion of the medial malleolus.
Changes in muscle contractile characteristics (with tensiomyography (TMG)) | Baseline and after 4 weeks
  Muscle involuntary contractile characteristics of the lower-limb muscles-the rectus femoris (RF), vastus medialis (VM), vastus lateralis (VL), biceps femoris (BF), semitendinosus (ST), tibialis anterior (TA), gastrocnemius medialis (GM) and gastrocnemius lateralis (GL)-will be recorded by measuring the response of these muscles to an induced electric stimulus (provoked by two self-adhesive electrodes) using TMG equipment on both the left and right lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Dovile Kiele, PhD, Principal Investigator — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania